CLINICAL TRIAL: NCT06230744
Title: A Novel Intervention for Weight Loss in Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Northwestern University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB23-1677; 1R01DK136214-01A1 (NIH)
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Other): Diet and exercise coaching
  Interventions: Behavioral: Lifestyle
- Lifestyle Intervention II (Experimental): Diet and exercise coaching
  Interventions: Behavioral: Lifestyle II

INTERVENTIONS:
Behavioral: Lifestyle — All participants will receive diet and exercise goals and coaching.
  Arms: Lifestyle Intervention
Behavioral: Lifestyle II — All participants will receive diet and exercise goals and coaching.
  Arms: Lifestyle Intervention II

SUMMARY:
Obesity and cardiometabolic risks are significant public health issues, with about two-thirds of U.S. adults overweight or obese. Weight loss can prevent these health problems, but current lifestyle interventions have limited success. New, effective strategies are needed to address this rising issue at the population level. The goal of this clinical trial is to investigate how a behavioral intervention combined with technology impacts weight loss in young adults. The main questions it aims to answer are:

• How does the combination of behavioral intervention and technology influence weight loss in young adults?

DETAILED DESCRIPTION:
The study team is seeking volunteers to participate in a research study to help better understand how a behavioral intervention combined with technology may impact weight loss. Participation will span approximately 6 months. Participants will be required to attend up to 5 visits at the University of Chicago. Those visits will include daytime visits to a clinic involving fasted blood draws and completion of surveys. During the study, participants will regularly record their weight using a digital scale, input their daily food intake into a smartphone app, and wear a wrist activity monitor to track their physical activity. Participants will also be paired with a trained coach to guide and assist their progress over their 6 months of participation.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (BMI 25.5- 34.9 kg/m2) men and women
* Ages 18 to 40 years
* Weight stable (no change >25 lbs in the past 3 months)
* Owns a smartphone and willing to install the study app

Exclusion Criteria:

* Presence of obstructive sleep apnea or history of any other sleep disorder.
* Irregular menses, menopausal symptoms or post-menopausal, currently pregnant, trying to get pregnant or nursing
* Regular travel across time zones
* Subjects who are currently following a weight loss regimen or any other special diet or exercise programs
* Increased fractional lean body mass (e.g., athletes)
* Unable to walk, using an assistive device for mobility, or any contraindications to exercise
* Diabetes
* Claustrophobia
* Excessive alcohol (>2 drinks/day) or caffeine (>300mg/day) intake, regular nicotine use, substance abuse.
* Abnormal findings on screening blood testing.
* Participants taking any prescription, over-the-counter drugs/supplements that can affect sleep or weight.
* Major psychiatric or any eating disorder, and any acute or chronic medical condition that increase the risk of interventions (e.g., heart disease)
* Any underlying disease likely to limit life span and/or increase risk of interventions including cardiovascular disease (e.g. unstable angina, heart failure requiring hospitalization in the past 6 months, significant heart block or arrhythmias, NYHA Class>2), pulmonary disease with dependence on oxygen or daily use of bronchodilators, cancer requiring treatment in the past 5 years unless the prognosis is considered good, active or chronic infection, thyroid disease and other endocrine disorders (e.g. Cushing syndrome, acromegaly), hepatitis or other chronic gastrointestinal disease (pancreatitis, inflammatory bowel disease), renal disease, significant anemia, recent surgery or significant abdominal surgery, major psychiatric or any eating disorder, acute coronary syndrome or stroke in the past 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | Baseline and 6 months
  Change in weight [kg] at 6 months. Weight will be measured by research staff during each visit in the morning in duplicate in the fasted state after voiding using calibrated digital scales, wearing a hospital gown.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tasali, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States